CLINICAL TRIAL: NCT02155439
Title: Treatment of Keloidscars With Intralesional Triamcinolone and 5-fluorouracil Injections-prospective, Randomized, Controlled Trial - Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Kristiina Hietanen, MD, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 140260M; 2013-004512-22 (EudraCT Number)
Record Dates: First submitted 2014-04-09; First posted 2014-06-04 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Keloidscars
Keywords: Prospective, randomized controlled trial - pilot study
MeSH Terms: interventions — Fluorouracil; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triamcinolone (Active Comparator): kortikosteroid
  Interventions: Drug: 5-fluorouracil
- 5-fluorouracil (Active Comparator): antimitotic drug
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: 5-fluorouracil — antimitotic drug
  Other Names: Fluorouracil Accord
  Arms: Triamcinolone
Drug: Triamcinolone
  Other Names: Lederspan
  Arms: 5-fluorouracil

SUMMARY:
The aim of study is examine the efficacy of intralesional 5-fluorouracil injections in keloid disease treatment.

ELIGIBILITY:
Inclusion Criteria:

* Person who has a keloidscar which could be treated with injection treatment

Exclusion Criteria:

* Pregnancy, lactating, renal or liver failure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Symptoms (pain, itching) of keloids and appearance of keloid | baseline and one year
  Change from baseline symptoms of scars baseline at one year with POSAS score

SECONDARY OUTCOMES:
Concentration change of hemoglobin and melanin | 0 week, 3 week, 6 week, 12 week, 1 year
  Camera analysis with spectrocutometry

OTHER OUTCOMES:
Inflammatory cells and their different populations, blood vessel density, fibroplast proliferation (KI67) and estrogenreseptor | 0 week, 3 week, 6 week, 12 week, 1 year
  immonuhistochemical analysis with punch biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere university hospital, Tampere, Finland